CLINICAL TRIAL: NCT03195530
Title: Bispectral Index (BIS) Values Required for an Adequate Depth of Anesthesia in Elderly Patients Using Propofol, According to the Characteristic Electroencephalographic Pattern
Brief Title: Bispectral Index (BIS) Values Required for an Adequate Depth of Anesthesia in Elderly Patients Using Propofol
Status: Terminated | Type: Observational
Why Stopped: Out of funding, no differences between groups
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 161207002
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients: Patients over 65 years, scheduled to general surgery, requiring general anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Induction of anesthesia using propofol, and recording the BIS values and EEG patterns during the induction

SUMMARY:
A correlation between the bispectral index values and electroencephalographic patterns at the loss of consciousness (LOC) when using propofol in elderly patients, has not been determined.

Our aim is to describe the BIS values and the power of the alpha band in the electroencephalography in elderly patients, at the LOC moment.

DETAILED DESCRIPTION:
Propofol is an anesthetic drug regularly used in elderly patients requiring anesthesia. The electroencephalographic pattern recognized when propofol is administered, is different to the pattern obtained in younger patients. Both groups presents an alpha and slow bands, but they differ in the intensity of the signal. Younger patients presents more intense electroencephalographic bands than older patients.

Bispectral index (BIS) is a clinical indicator used to evaluate the depth of anesthesia. A correlation between this indicator and the power of electroencephalographic bands has not been determined.

We will describe the LOC moment of elderly patients receiving propofol as anesthetic for general surgery, with the EEG characteristic bands and the BIS value obtained at that moment. The BIS values related to the EEG characteristic bands can be described, to correlate the actual indicators of depth of anesthesia with new parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years
* Scheduled for elective surgery requiring general anesthesia
* American Society of Anesthesiology (ASA) Score I or II

Exclusion Criteria:

* Patients with neurological diseases
* Requiring the use of two or more drugs affecting Central nervous system
* History of drugs or alcohol abuse
* Body mass index over 35 kg/m^2
* Propofol allergy
* Cardiac congestive failure
* History of coronary syndrome
* Minimental test altered (Score under 24 points)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients scheduled for surgery are an understudied population. Incidence of postoperative delirium and other complications can be related to changes in cerebral dynamics under anesthesia, with effects observed even after the use of anesthetics agents.
  To characterize changes in EEG patterns under the induction of anesthesia, can give new information to understand the physiology of the elderly brain under anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
BIS values at which EEG patterns (Slow and alpha bands) appears in elderly population using propofol | Induction of anesthesia
  To describe the BIS values correlated to specific EEG patterns

SECONDARY OUTCOMES:
Propofol concentration required to observe specific EEG patterns | Induction of anesthesia
  To describe the serum propofol concentrations required for induction of anesthesia, to observe alpha and slow bands at the EEG.

CONTACTS AND LOCATIONS:
Locations (1):
- Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No